CLINICAL TRIAL: NCT02673411
Title: Diagnostic Performance of Shear Wave Elastography for Fibrosis Evaluation: Preliminary Study
Brief Title: Ultrasonography SWE for Hepatic Fibrosis Evaluation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH-2016-0065
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cirrhosis
Keywords: elastography; ultrasonography
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ultrasound shear wave elastography — ultrasound shear wave elastography is performed in GE ultrasound scanner according to guidelines of ultrasound elastography.
  Other Names: GE LOGIQ E9

SUMMARY:
The purpose of this study is to measure diagnostic performance of ultrasound shear wave elastography to detect advanced hepatic fibrosis.

DETAILED DESCRIPTION:
Hepatic fibrosis causes liver dysfunction and HCC. Since hepatic fibrosis is reversible dynamic condition, its monitoring is important to predict long term outcome and to determine treatment plan.

The reference of standard to diagnose hepatic fibrosis is biopsy, but recently non-invasive method such as stiffness imaging has been drawing a lot of attention. In this study, ultrasound shear wave elastography will be performed and its diagnostic performance to detect advanced hepatic fibrosis (= > F2) will be measured using histologic grade as a reference.

ELIGIBILITY:
Inclusion Criteria:

* volunteers who agree to undergo US shear elastography OR
* patients with chronic liver disease who are scheduled to undergo liver resection or liver parenchymal biopsy.

AND

* = or > 18 years
* sign informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to undergo liver resection or liver biopsy (n=138). Volunteers who agree to undergo US shear wave elastography (n=20) to determine inter-observer agreement.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
diagnostic performance to detect advanced hepatic fibrosis | 1 month
  from ultrasound SWE to perform hepatic resection or percutaneous liver biopsy in patients (with histologic diagnosis)

SECONDARY OUTCOMES:
interobserver agreement of ultrasound SWE | 1 day
  two observers perform ultrasound SWE on the same day in volunteers.
agreement with MR elastography | 1 month
  interval between US and MR elastography in patients with available MR elastography
Technical success rate | 6 months
  technical success or failure of US elastography using GE LOGIQ E9 scanner in ALL study population
Reliable measurement rate | 6 months
  reliable measurement rate (interquartile range of serial measurement/median LS value <30%) in patients with technically successful US elastography

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No